CLINICAL TRIAL: NCT04956510
Title: Investigation of Individuals With Osteoarthritis in Terms of ICF Components Based of ICF Comprehensive Core Set for Osteoarthritis and Quality of Life
Brief Title: Osteoarthritis in Terms of ICF Components
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, MSc, PT, Research Assistant, Pamukkale University
Other Study IDs: PAU
Record Dates: First submitted 2021-07-02; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis; Quality of Life; OUTCOME MEASURES
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation — health status and quality of life were evaluated

SUMMARY:
Osteoarthritis (OA) is a common degenerative disease associated with functional impairments, activity limitations, participation restrictions, as well as poor quality life. Therefore, the comprehensive assessment is important to determine how complex problems affect patients with OA. The first aim of this study was to link and allocate items of The Western Ontario and McMaster Universities (WOMAC) OA index with ICF Comprehensive Core Set for osteoarthritis. The second aim was to examine the relationship between the quality of life and each ICF component's scores determined based on clinical data of WOMAC in OA.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with OA according to American College of Rheumatology clinical criteria for OA of the knee or hip;[14,15]
* being in the age range 18-65; and
* absence of other diseases affecting functions and daily life (orthopedic, neurological, cardiovascular, metabolic disease and lung pathology).

Exclusion Criteria:

* comorbidity affecting lower extremity and functions (patellofemoral pain syndrome, rheumatoid arthritis, ligament tear, meniscus);
* previous lower extremity surgery;
* Intra-articular steroid or hyaluronic acid injection in the last three months
* cognitive impairments;
* pregnancy; and
* illiteracy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty-seven patients with OA were included in this study, who met inclusion criteria and were diagnosed with OA by the same rheumatologist according to the American College of Rheumatology Clinical Classification Criteria for OA.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities (WOMAC) OA Index: | 15 min
  The WOMAC Index is a self-administered, disease-specific questionnaire consisting of 24 items which are widely used in the evaluation of hip and knee OA. It consists of 24 items: pain (5 items), stiffness (2 items), and physical function (17 items). High score indicates worse pain, stiffness, and functional limitations.
Nottingham Health Profile (NHP): | 15 min
  NHP is a widely used measure of perceived distress of patients in physical, emotional and social domains. It consists of 38 items which are physical mobility (8 items), pain (8 items), sleep (5 items), emotional reactions (9 items), social isolation (5 items) and energy level (3 items). Questions have "yes" or "no" answers. Higher score indicates greater distress

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University School of Physical Therapy and Rehabilitation, Denizli, Turkey (Türkiye)